CLINICAL TRIAL: NCT06644534
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral TTI-0102 for Treatment of Patients With Mitochondrial Encephalomyopathy, Lactic Acidosis and Stroke-like Episodes (MELAS)
Brief Title: A Study to Assess TTI-0102 vs Placebo in MELAS Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thiogenesis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTI-MITO-001
Record Dates: First submitted 2024-09-29; First posted 2024-10-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: MELAS Syndrome; Mitochondrial Encephalomyopathy, Lactic Acidosis and Stroke-like Episodes (MELAS)
MeSH Terms: conditions — MELAS Syndrome | interventions — cysteamine-pantetheine disulfide

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized, Double-Blind, Placebo-Controlled Twelve (12) patients will be randomized on a 2:1 (active:placebo) ratio, with 8 receiving TTI-0102 and 4 receiving a placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigator and sponsor will be blinded to active:placebo assignment and to PK measurements during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TTI-0102 (Experimental): cysteamine-pantetheine disulfide
  Interventions: Drug: TTI-0102
- Placebo (Placebo Comparator): Pearlitol® 100 SD (mannitol)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TTI-0102 — (cysteamine-pantetheine disulfide)
  Arms: TTI-0102
Drug: Placebo — Pearlitol® 100 SD (mannitol)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study. Prior to treatment, patients will undergo a screening visit. If eligible, each subject will return for a Day 1 visit and will receive their first dose of investigational product (TTI-0102 or placebo). At the end of the first week of treatment, subjects will return for a Week 1/Day 8 study visit to assess study drug dosing/tolerance and instruct on dosing for the upcoming second week of treatment.

For the first 8 weeks of treatment, subjects will alternate between returning to the clinic for detailed assessments (Weeks 4 and 8) and receiving a telephone call from the Investigator team to assess safety and TTI-0102 dose (Weeks 2 and 6) and the potential need for an immediate unscheduled study visit.

After the first 8 weeks of treatment, subjects will continue to return to the clinic for monthly assessments at Weeks 12, 16, 20. The Study Exit visit will occur at Week 24, and subjects will be offered to continue on an open-label extension study of TTI-0102. If a subject does not complete the study, they will be asked to return for a Study Exit visit 4 weeks after last study drug dose.

Primary Objective The primary objective of this study is to assess the efficacy, safety and tolerability of oral TTI 0102 compared to placebo, for up to 6 months in patients with MELAS.

Secondary Objective The secondary objectives of this study are to assess the efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of cysteamine after oral administration of TTI-0102 at steady state, in patients with MELAS on a stable dose of TTI-0102.

This is a randomized, double-blind, placebo-controlled study. Prior to treatment, patients will undergo a screening visit. If eligible, each subject will return for a Day 1 visit and will receive their first dose of investigational product (TTI-0102 or placebo). At the end of the first week of treatment, subjects will return for a Week 1/Day 8 study visit to assess study drug dosing/tolerance and instruct on dosing for the upcoming second week of treatment.

For the first 8 weeks of treatment, subjects will alternate between returning to the clinic for detailed assessments (Weeks 4 and 8) and receiving a telephone call from the Investigator team to assess safety and TTI-0102 dose (Weeks 2 and 6) and the potential need for an immediate unscheduled study visit.

After the first 8 weeks of treatment, subjects will continue to return to the clinic for monthly assessments at Weeks 12, 16, 20. The Study Exit visit will occur at Week 24, and subjects will be offered to continue on an open-label extension study of TTI-0102. If a subject does not complete the study, they will be asked to return for a Study Exit visit 4 weeks after last study drug dose.

Study Drug Dosing To prevent any manifestation of intolerance at the initiation of drug treatment, only half a dose (2.75 grams) will be given once a day for the first week of treatment. During the following weeks of treatment, patients will be given a full dose of 5.5 grams once a day.

Interim Data Review After nine (9) patients have completed three months of treatment (the Week 12 visit) an interim data cut will take place to assess safety and potential efficacy signals. Even if no indications of efficacy are detected at this early stage, the trial itself will not be terminated unless there is a serious safety concern (i.e., protocol-defined Stopping Criteria are met).

ELIGIBILITY:
Inclusion Criteria:

1. Patient or Patient's legally designated representative has given written informed consent before any study-related activities are carried out and is able to understand the full nature and purpose of the trial, including possible risks and adverse effects. Patient has provided assent according to local/institutional requirements.
2. Males and females between 16 and 60 years of age at screening.
3. Diagnosis of mitochondrial encephalomyopathy, lactic acidosis and stroke-like episodes (MELAS), defined as:

   - mtDNA mutation known to be associated with MELAS and MELAS phenotype (Emmanuele et al., 2022) including but not limited to: m.3243A>G, m.13513G>A, m.10191T>C, m. 3271T>C, m. 13136_15374del, m. 8363G>A. Mutation must have heteroplasmy >50% characterized by mutation load in urinary epithelium or blood.

   AND

   - two or more of the following clinical symptoms indicative of MELAS phenotype: diabetes, myopathy, seizures, at least one historic stroke-like episode, and exercise intolerance.
4. Moderate disease severity defined as Newcastle Mitochondrial Disease Adult Scale (NMDAS) score between 15 to 45 inclusive.
5. Able to complete a 12-minute walk test (12-MWT) distance of at least 150 meters and no more than 1000 meters within 30 days prior to, or at time of screening.
6. Subjects regularly taking dietary supplements including but not limited to creatine, alpha-lipoic acid, CoQ10, B vitamins, levocarnitine shall have been taking them for at least 3 months pre-study and will agree to continue taking them throughout the study (from the Screening Visit to Study Exit).
7. With respect to concomitant medications, the subject must:

   1. Be willing to abstain from initiating new dietary supplements and non-prescribed medications, except as permitted by the Investigator throughout the study.
   2. Be on a stable dose of medications prescribed for seizure management and prevention. Stable dose in this context means unchanged for at least 30 days prior to the Screening Visit.
8. Willing and able to comply with study drug dosing requirements, i.e., able to ingest study drug solution orally.
9. Female participants:

   * Must be of nonchildbearing potential (i.e., surgically sterilized [hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the screening visit]) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause, and a follicle-stimulating hormone [FSH] level >40 IU/L at the screening visit), or
   * If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to the use of acceptable forms of highly effective contraception (refer to protocol Section 19.2) from the time of signing the consent form until at least 30 days after the last dose of the study drug.
10. Male participants:

    * Engaging in any sexual intercourse, including those who are infertile and do not produce sperm (e.g. post-vasectomy), must abstain from unprotected sex until the Study Exit visit.
    * Must agree to abstain from sperm donation, and if engaging in sexual intercourse with a female of child bearing potential must agree to the use of an acceptable form of highly effective contraception (refer to protocol Section 19.2) from the time of signing the consent form until at least 30 days after the last dose of study drug.
11. Have suitable venous access for blood sampling.
12. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. Documented diagnosis of concurrent inborn errors of metabolism.
2. Non-elective hospitalization related to their mitochondrial disease or direct complication of disease within 60 days prior to the Screening Visit.
3. Overt comorbidity preventing them from safely performing an exercise. In particular, patients suffering from cardiovascular, neurological disorders (e.g. ataxia, sequel blindness from pseudostroke, peripheral neuropathy) or advanced osteo-arthrosis.
4. Treatment with taurine during the previous month, and not willing to discontinue for the duration of the trial.
5. Platelet count, lymphocyte count or hemoglobin level below the lower limit of normal (LLN) at screening.
6. Hepatic insufficiency with liver enzyme tests (alkaline phosphatase, AST or ALT) greater than 2.5 times to upper limit of normal (ULN) at screening.
7. Bilirubin > 1.2 g/dL at screening.
8. Renal insufficiency, defined as 1) a requirement for chronic dialysis or 2) serum creatinine ≥1.2 mg/dl or creatinine clearance <60 ml/min
9. Severe gastrointestinal disease including gastroparesis.
10. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs. Examples: malabsorption requiring TPN, chronic diarrhea, bouts of pseudo obstruction.
11. Severe end-organ hypo-perfusion syndrome secondary to cardiac failure resulting in lactic acidosis.
12. Patients with suspected elevated intracranial pressure, pseudotumor cerebri (PTC) and/or papilledema.
13. History of angina, myocardial infarction, or cardiac surgery within 2 years prior to screening.
14. History of drug or alcohol abuse.
15. History of pancreatitis.
16. Known or suspected hypersensitivity to cysteamine.
17. Allergy to any medicine containing mercaptamine, penicillamine or known hypersensitivity to any of the study drug ingredients.
18. Evidence of or verbal attestation of Helicobacter pylori infection, presently, or within the last 90 days prior to Screening.
19. Use of any live vaccinations within 30 days prior to the first study drug administration except for the influenza vaccine (note that COVID-19 vaccine is permitted).
20. For women of childbearing potential, a positive urine pregnancy test and confirmatory positive serum test at screening. Must not be currently breastfeeding.
21. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
22. Participation in another investigational clinical trial within 30 days if a drug, or 90 days for a biologic or device, prior to screening.
23. Any other condition or prior therapy that in the opinion of the Investigator would make the subject unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Change in functional capacity | Day 1/Baseline to Week 24/Study Exit
  12-minute walking test (12-MWT)
Safety and Tolerability: Incidence of Treatment-Emergent Adverse Events | Day 1/Baseline to Week 24/Study Exit
  Adverse Events

SECONDARY OUTCOMES:
Efficacy: Fatigue | Day 1/Baseline to Week 24/Study Exit
  Fatigue Severity Scale (FSS)
Efficacy: Quality of Life (QoL) | Day 1/Baseline to Week 24/Study Exit
  Qualify of Life (WHOQOL-BREF)
Pharmacokinetic parameter: Cmax | Day 1/Baseline to Week 24/Study Exit
  cysteamine in plasma
  cysteamine, pantothenic acid (vitamin B5) and taurine
Pharmacokinetic parameter: Tmax | Day 1/Baseline to Week 24/Study Exit
  cysteamine in plasma
Pharmacokinetic parameter: AUC | Day 1/Baseline to Week 24/Study Exit
  cysteamine in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P Rioux, MD, PhD, Study Director — Thiogenesis Therapeutics, Inc.
Locations (2):
- Angers University Hospital Center (CHU Angers), Angers, France
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No